CLINICAL TRIAL: NCT00342654
Title: Nutritional Intervention Trials in Linxian China- Continued Follow-up
Brief Title: Nutrition Intervention Trials in Linxian Follow-up Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999031; OH99-C-N031
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Epidemiology; Cancer; Environment; Genetics; Nutrition; Natural History
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants from two large, nutritional intervention trials that were conducted in Linxian, China between 1985-1991.

SUMMARY:
Two large, nutritional intervention trials were conducted in Linxian, China between 1985-1991. These trials tested the effect of multiple vitamins and minerals in the prevention of esophageal cancer in a population with the highest known rate for this disease in the world. Results from the trials showed that Beta-carotene + Vitamin E + selenium reduced total mortality, total cancer mortality, and stomach cancer incidence and mortality. Multivitamins/minerals also showed reduction in premalignant lesions. Preliminary follow-up data obtained for the time period after cessation of intervention in 1991 suggests that the observed benefit for total and cancer mortality is reduced but that the benefit for stomach cancer remains.

The objectives of the follow-up study are: (1) to continue to determine cancer incidence and all causes of mortality in trial participants after intervention to permit examination of potential effects of the interventions on total and cause-specific mortality and cancer incidence in the post-intervention period; (2) to conduct a cross-sectional nutritional survey in a subsample of living trial participants to evaluate their nutritional status, asses the validity of dietary questionnaires, and relate neurologic status to vitamin B12 plasma levels; (3) to collect a blood sample from all living trial participants to permit further etiologic investigations of genetic and environmental hypotheses; and (4) to perform nested case-control studies of selected genetic and environmental hypotheses.

To accomplish the objectives of the follow-up study, we will: (1) determine updated vital status and cancer status data on all trial participants via monthly checks of village doctor records and quarterly checks of the Linxian Cancer Registry; conduct a Vital/Cancer Status Interview Survey among all (n-34,000 trial participants (or their surrogates); identify, collect, and store all available diagnostic materials for trial participants identified as having developed cancer or died with cancer during the follow-up period; (2) conduct a Nutritional Survey on a subsample (n-1000) of living trial participants that will include (a) a physical exam and brief medical history, (b) a neurologic history, (c) a cognitive function exam, (d) a hair/mouth skin exam, (e) a neurological exam, (f) a nutritional questionnaire, and (g) collection of a blood sample for hematologic/biochemical analyses; (3) conduct a Blood Collection Survey of all living trial participants (n-23,000) to obtain (a) a physical exam and brief medical history and (b) a single 10-ml blood sample for separation and preservation as WBCs (both viable and nonviable), RBCs, and plasma for genetic (e.g., xenobiotic polymorphisms) and environmental (e.g., plasma ascorbic acid) hypothesis testing; and (4) perform Nested Case-Control Studies of selected genetic and environmental hypothesis related to the etiology and prevention of esophageal cancer and stroke. These will be done using serum from the new cancer and stroke cases (-2500) and controls (-2500) previously identified from 1991-1996, as well as using new cancer and stroke cases and controls for the period 1996-2004 (-9000).

The followup for endpoints will continue monthly for an additional 5 years (through the year 2003). The Nutritional Survey and Blood Collection Survey will be conducted in the spring of 1999. The Nested Case-Control studies will be performed annually beginning in 2000, and the Vital/Cancer Interview Survey will be conducted in the Spring of 2001.

DETAILED DESCRIPTION:
Two large, nutritional intervention trials were conducted in Linxian, China between 1985-1991. These trials tested the effect of multiple vitamins and minerals in the prevention of esophageal cancer in a population with the highest known rate for this disease in the world. Results from the trials showed that Beta-carotene + Vitamin E + selenium reduced total mortality, total cancer mortality, and stomach cancer incidence and mortality. Multivitamins/minerals also showed reduction in premalignant lesions. Preliminary follow-up data obtained for the time period after cessation of intervention in 1991 suggests that the observed benefit for total and cancer mortality is reduced but that the benefit for stomach cancer remains.

The objectives of the follow-up study are: (1) to continue to determine cancer incidence and all causes of mortality in trial participants after intervention to permit examination of potential effects of the interventions on total and cause-specific mortality and cancer incidence in the post-intervention period; (2) to conduct a cross-sectional nutritional survey in a subsample of living trial participants to evaluate their nutritional status, asses the validity of dietary questionnaires, and relate neurologic status to vitamin B12 plasma levels; (3) to collect a blood sample from all living trial participants to permit further etiologic investigations of genetic and environmental hypotheses; and (4) to perform nested case-control studies of selected genetic and environmental hypotheses.

To accomplish the objectives of the follow-up study, we will: (1) determine updated vital status and cancer status data on all trial participants via monthly checks of village doctor records and quarterly checks of the Linxian Cancer Registry; conduct a Vital/Cancer Status Interview Survey among all (n approximately 34,000 trial participants (or their surrogates); identify, collect, and store all available diagnostic materials for trial participants identified as having developed cancer or died with cancer during the follow-up period; (2) conduct a Nutritional Survey on a subsample (n approximately 1000) of living trial participants that will include (a) a physical exam and brief medical history, (b) a neurologic history, (c) a cognitive function exam, (d) a hair/mouth skin exam, (e) a neurological exam, (f) a nutritional questionnaire, and (g) collection of a blood sample for hematologic/ biochemical analyses; (3) conduct a Blood Collection Survey of all living trial participants (n approximately 23,000) to obtain (a) a physical exam and brief medical history and (b) a single 10-ml blood sample for separation and preservation as WBCs (both viable and nonviable), RBCs, and plasma for genetic (e.g., xenobiotic polymorphisms) and environmental (e.g., plasma ascorbic acid) hypothesis testing; and (4) perform Nested Case-Control Studies of selected genetic and environmental hypothesis related to the etiology and prevention of esophageal cancer and stroke. These will be done using serum from the new cancer and stroke cases (approximately 2500) and controls (approximately 2500) previously identified from 1991-1996, as well as using new cancer and stroke cases and controls for the period 1996-2004 (approximately 9000).

The followup for endpoints will continue monthly for an additional 5 years (through the year 2003). The Nutritional Survey and Blood Collection Survey will be conducted in the spring of 1999. The Nested Case-Control studies will be performed annually beginning in 2000, and the Vital/Cancer Interview Survey will be conducted in the Spring of 2001.

ELIGIBILITY:
* No eligibility criteria listed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from two large, nutritional intervention trials that were conducted in Linxian, China between 1985-1991. These trials tested the effect of multiple vitamins and minerals in the prevention of esophageal cancer in a population with the highest known rate for this disease in the world.
Sampling Method: Non-Probability Sample
Enrollment: 32902 (Actual)
Dates: Start 1999-05-20 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Determine cancer incidence and all causes of mortality in trial participants in the post-intervention period and conduct studies ofselected genetic and environmental hypotheses related to the etiology and prevention of esophageal cancer and s... | Ongoing
  analysis is ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Murphy G, Freedman ND, Michel A, Fan JH, Taylor PR, Pawlita M, Qiao YL, Zhang H, Yu K, Abnet CC, Dawsey SM. Prospective study of Helicobacter pylori antigens and gastric noncardia cancer risk in the nutrition intervention trial cohort. Int J Cancer. 2015 Oct 15;137(8):1938-46. doi: 10.1002/ijc.29543. Epub 2015 May 5. PMID 25845708
- [Background] Abnet CC, Freedman ND, Hu N, Wang Z, Yu K, Shu XO, Yuan JM, Zheng W, Dawsey SM, Dong LM, Lee MP, Ding T, Qiao YL, Gao YT, Koh WP, Xiang YB, Tang ZZ, Fan JH, Wang C, Wheeler W, Gail MH, Yeager M, Yuenger J, Hutchinson A, Jacobs KB, Giffen CA, Burdett L, Fraumeni JF Jr, Tucker MA, Chow WH, Goldstein AM, Chanock SJ, Taylor PR. A shared susceptibility locus in PLCE1 at 10q23 for gastric adenocarcinoma and esophageal squamous cell carcinoma. Nat Genet. 2010 Sep;42(9):764-7. doi: 10.1038/ng.649. Epub 2010 Aug 22. PMID 20729852
- [Background] Qiao YL, Dawsey SM, Kamangar F, Fan JH, Abnet CC, Sun XD, Johnson LL, Gail MH, Dong ZW, Yu B, Mark SD, Taylor PR. Total and cancer mortality after supplementation with vitamins and minerals: follow-up of the Linxian General Population Nutrition Intervention Trial. J Natl Cancer Inst. 2009 Apr 1;101(7):507-18. doi: 10.1093/jnci/djp037. Epub 2009 Mar 24. PMID 19318634
- [Derived] Yang H, Wang J, Wang X, Sun W, Tong C, Fan J, Qiao Y, Abnet CC. Weight change and all-cause and cause-specific mortality: A 25-year follow-up study. Chin Med J (Engl). 2024 May 20;137(10):1169-1178. doi: 10.1097/CM9.0000000000002970. Epub 2024 Jan 29. PMID 38282387
- [Derived] Yang H, Wang JB, Wang XK, Fan JH, Qiao YL. Association between type of drinking water and upper gastrointestinal cancer incidence in the Linxian General Population. BMC Cancer. 2023 May 4;23(1):397. doi: 10.1186/s12885-023-10887-2. PMID 37142988
- [Derived] Fan JH, Wang JB, Wang SM, Abnet CC, Qiao YL, Taylor PR. Longitudinal change in blood pressure is associated with cardiovascular disease mortality in a Chinese cohort. Heart. 2018 Nov;104(21):1764-1771. doi: 10.1136/heartjnl-2017-312850. Epub 2018 Apr 24. PMID 29691288
- [Derived] Wang SM, Taylor PR, Fan JH, Pfeiffer RM, Gail MH, Liang H, Murphy GA, Dawsey SM, Qiao YL, Abnet CC. Effects of Nutrition Intervention on Total and Cancer Mortality: 25-Year Post-trial Follow-up of the 5.25-Year Linxian Nutrition Intervention Trial. J Natl Cancer Inst. 2018 Nov 1;110(11):1229-1238. doi: 10.1093/jnci/djy043. PMID 29617851
- [Derived] Fan JH, Wang JB, Wang SM, Abnet CC, Qiao YL, Taylor PR. Body mass index and risk of gastric cancer: A 30-year follow-up study in the Linxian general population trial cohort. Cancer Sci. 2017 Aug;108(8):1667-1672. doi: 10.1111/cas.13292. Epub 2017 Jun 30. PMID 28594442
- [Derived] Chen W, Wang JB, Abnet CC, Dawsey SM, Fan JH, Yin LY, Yin J, Taylor PR, Qiao YL, Freedman ND. Association between C-reactive protein, incident liver cancer, and chronic liver disease mortality in the Linxian Nutrition Intervention Trials: a nested case-control study. Cancer Epidemiol Biomarkers Prev. 2015 Feb;24(2):386-92. doi: 10.1158/1055-9965.EPI-14-1038. Epub 2015 Jan 22. PMID 25613115
- [Derived] Wang JB, Abnet CC, Fan JH, Qiao YL, Taylor PR. The randomized Linxian Dysplasia Nutrition Intervention Trial after 26 years of follow-up: no effect of multivitamin supplementation on mortality. JAMA Intern Med. 2013 Jul 8;173(13):1259-61. doi: 10.1001/jamainternmed.2013.6066. No abstract available. PMID 23712839